CLINICAL TRIAL: NCT04436445
Title: Effect of Neurogenic Acupoint Cupping on Hs-CRP and Pain Perception in Women With Chronic Pevic Pain
Brief Title: Effect of Neurogenic Acupoint CUPPING ON WOMEN WITH CHRONIC PELVIC PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, Rehab Tareq Mohamad, physiotherapist in Ministry of Health and Population, Egypt, Ministry of Health and Population, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO:P.T.REC/012/002019
Record Dates: First submitted 2020-06-02; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Chronic Pelvic Pain
Keywords: chronic pelvic pain; dry cupping; neurogenic acupoint

STUDY DESIGN:
Intervention Model Description: women's with chronic pelvic pain
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- dry cupping (Active Comparator): Dry cupping is considered to be a noninvasive and inexpensive technique, used worldwide to treating patients with pain syndromes It is in fact a type of physical therapy which is applied by the specialists of acupuncture or other individuals. It improves the subcutaneous blood flow and, as a result, stimulates the autonomic nervous system and reduces the pai
  Interventions: Combination Product: dry cupping
- Life style modification (Active Comparator): lifestyle modifications in the form of dietary recommendations, exercises and sleep quality improvement for 8 weeks.The life style modification followed in the treatment: Avoid consumption of all kinds of alcohol beverages. Avoid consumption of spicy foods, pepper, chili and coffee Follow a correct diet assuming each day 50% carbohydrates,30% fats and 20% proteins Increase your intake of fruits, vegetables and foods rich of natural fibers (dark bred, vegetables, spinaches).
  8 hour sleep at night 40 minutes of walking 3time per week.
  Interventions: Other: Life style modification

INTERVENTIONS:
Combination Product: dry cupping — represents the location and clinical importance of each acupoint. First, the position of the patient will be supine lying for SP6, SP9, KI6, GB34 and CV6 acupoints and it will be prone lying for B23 acupoint. Second, the skin will be cleaned by alcohol then cups will be placed on the acupoints. Dry cupping for SP6, SP9, KI6 and GB34 acupoints will be applied using small cups while dry cupping for CV6 and B23 will be applied using large cups. Third, a negative pressure will be applied with a manual handle. Finally, the cups will be removed after 5 to 15 minutes by pressing one side of the skin with a finger to release the vacuum slowly.
  Arms: dry cupping
Other: Life style modification — Life style modification
  Arms: Life style modification

SUMMARY:
PURPOSE:

The purpose of this study is to determine the effect of dry cupping on women with chronic pelvic pain.

BACKGROUND:

Recent studies have examined the efficacy of dry cupping on acupoints for various pain-related conditions. They showed good result . However, no studies up to date has been evaluated the effect of dry cupping in treating Chronic pelvic pain. Therefore, this study is the first one which aims to investigate the effect of dry cupping on women suffering from Chronic pelvic pain. This study may expand the role of physiotherapy in woman's health.

HYPOTHESE:

There is no effect of bioptron light therapy on postmenopausal osteoporosis.

RESEARCH QUESTION:

There is no effect of dry cupping on chronic pelvic pain.

DETAILED DESCRIPTION:
Chronic pelvic pain is a highly prevalent debilitating disease with negative impact on the quality of life and productivity of women. The estimated prevalence of CPP is 3.8% among women aged 15-73 years, ranging from 14% to 24% among women of reproductive age, with a direct impact on their marital, social and professional life .

A specific diagnosis for CPP is often difficult; no diagnosis is made in 60% of patients . Treatment of these patients remains a challenge due to the diverse clinical signs and phenotypes. Several non-surgical as well as surgical strategies exist. However, many of the therapy approaches seem to have only limited effect in managing CPP . Additionally, many of the recommended medical and surgical interventions have a potential for harm in a proportion of women . Accordingly, an alternative therapeutic approach is desirable.

Dry cupping is considered to be a noninvasive and inexpensive technique, used worldwide to treating patients with pain syndromes . It is in fact a type of physical therapy which is applied by the specialists of acupuncture or other individuals. It improves the subcutaneous blood flow and, as a result, stimulates the autonomic nervous system and reduces the pain . The application of suction on selected acupoints produces hyperemia or hemostasis, which may result in a therapeutic effect .When compared to acupuncture, cupping therapy is a non-invasive therapy with relatively shorter treatment duration and less treatment cost .

Recent studies have examined the efficacy of dry cupping on acupoints for various pain-related conditions. They showed good results . However, no studies up to date has been evaluated the effect of dry cupping in treating CPP. Therefore, this study is the first one which aims to investigate the effect of dry cupping on women suffering from CPP. This study may expand the role of physiotherapy in woman's health

ELIGIBILITY:
Inclusion Criteria:

* thirty married women suffering from chronic pelvic pain
* Their age will range from 25 to 40 years old.
* Their BMI will be ≤ 30 kg/m2.
* They should be non-smokers.
* They should have sedentary life style without participation at any exercise training program during this study.
* Maximum parity number is three.
* Their score is less than 6 on The Interstitial Cystitis Symptom Index and Problem Index" (The O'Leary-Sant), to exclude Interstitial Cystitis.
* Their score on visual analog scale above 5.
* Their muscle strength is good in hip abductor, adductor, external rotator and internal rotator muscles .
* Their pelvic floor muscle strength is good.

Exclusion Criteria:

* Women having any serious physical disorders such as vertebral fractures, disk hernia, acute inflammation and deep venous thrombosis.
* Women having any problems in the acupoints such as fractures, ulcers, varicose veins, skin disease or inflammation.
* Women having history of cancer or congenital anomaly.
* Use of any kind of analgesic medications or contraceptive pills.
* Diabetic or hypertensive patient.
* Have any auto immune disease (rheumatoid, lupus), chest disease and cardiac disease.
* HS-CRP test exclusion patient during menses, patient suffering any medical condition increase inflammation ex cough, sneezing.
* Patient suffering from chronic pelvic pain due to another cause except PID.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
High sensitive C - reactive protein (Hs-CRP) | 8 weeks
Short-Form McGill Pain Questionnaire (SF-MPQ) | 8 weeks
  It is a reliable and valid instrument that is easier and quicker to use in clinical research than the McGill pain questionnaire (MPQ). It will be used to evaluate pain intensity for each woman in both groups before and after the end of treatment program. It consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Pelvic Pain Impact Questionnaire (PPIQ) | 8 weeks
  a questionnaire that assesses the impact of pelvic pain on women, that has high utility, sound psychometric performance, easy scoring, and high reliability, 10-item questionnaire consisted of 8 Likert questions and 2 supplemental, nonscored questions, the questionnaire targeted the pelvic pain population well, had appropriate Likert categories, constituted a unidimensional scale, and showed internal consistency. Test-retest reliability was highPelvic Pain Impact Questionnaire assesses the life impact of pelvic pain. It uses patient-generated language, is easily administered and scored, has very strong psychometric properties, and it is suitable for research and clinical settings across primary, secondary, and tertiary care

CONTACTS AND LOCATIONS:
Locations (1):
- They will be selected from 6th District Family Medicine Unit, Giza., Giza, Egypt